CLINICAL TRIAL: NCT06650124
Title: Induction of Remission in Autoimmune Hepatitis With Azathioprine vs. MMF
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12/8/2023-ACAD/E-12745/992
Record Dates: First submitted 2024-10-17; First posted 2024-10-21 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: Autoimmune Hepatitis
Keywords: utoimmune Hepatitis (AIH); Azathioprine (AZA); Mycophenolate Mofetil (MMF); Induction of Remission
MeSH Terms: conditions — Hepatitis, Autoimmune | interventions — Mycophenolic Acid; Azathioprine; Prednisolone

STUDY DESIGN:
Intervention Model Description: nterventional Study Model: Parallel Assignment Study Type: Interventional (Clinical Trial) Study Model: Parallel Assignment - Participants are randomly assigned to one of two groups (either receiving azathioprine or mycophenolate mofetil) and remain in their assigned group for the entire study.
  Masking: Double-blind (both participants and investigators are unaware of which treatment is being administered to prevent bias).
  Allocation: Randomized - Patients are randomly allocated to one of the two treatment groups.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Azathioprine + Prednisolone Arm (Active Comparator): Azathioprine + Prednisolone Arm Participants will receive azathioprine (AZA) in combination with prednisolone as part of their treatment regimen.
  Interventions: Drug: Azathioprine + Prednisolone
- Mycophenolate Mofetil + Prednisolone Arm (Active Comparator): Mycophenolate Mofetil + Prednisolone Arm Participants will receive mycophenolate mofetil (MMF) in combination with prednisolone as part of their treatment regimen.
  Interventions: Drug: Mycophenolate Mofetil + Prednisolone Participants will receive mycophenolate mofetil in combination.

INTERVENTIONS:
Drug: Mycophenolate Mofetil + Prednisolone Participants will receive mycophenolate mofetil in combination. — Participants in this arm will receive mycophenolate mofetil (MMF) starting at 1,000 mg/day for the first two weeks, increasing to 2,000 mg/day thereafter. This will be combined with prednisolone, beginning at 40-60 mg/day, with a tapering dose to 5-10 mg/day after 4-8 weeks, depending on the patient's response. MMF works by inhibiting inosine monophosphate dehydrogenase, which decreases lymphocyte proliferation, thereby reducing immune-mediated liver damage in autoimmune hepatitis. Prednisolone, a corticosteroid, is included to control inflammation during the induction phase of treatment. This intervention lasts for 24 weeks, with monitoring for biochemical remission (normalization of liver enzymes and IgG levels) and adverse events to assess the treatment's safety and efficacy.
  Arms: Mycophenolate Mofetil + Prednisolone Arm
Drug: Azathioprine + Prednisolone — In this arm, participants will receive azathioprine (AZA) starting at 50 mg/day for the first two weeks, followed by an increase to 100 mg/day. This dose will be combined with prednisolone, starting at 40-60 mg/day, with the dosage tapering to 5-10 mg/day after 4-8 weeks, depending on patient response. Azathioprine works as an immunosuppressive agent by inhibiting DNA synthesis in rapidly dividing immune cells, thereby reducing liver inflammation in autoimmune hepatitis. Prednisolone, a corticosteroid, is included to control inflammation during the initial treatment phase. The intervention lasts for 24 weeks with regular monitoring for biochemical remission, defined as normalization of liver enzymes (AST, ALT) and IgG levels, as well as the occurrence of adverse events to assess safety and tolerability.
  Arms: Azathioprine + Prednisolone Arm

SUMMARY:
The goal of this clinical trial is to determine the effectiveness of azathioprine (AZA) versus mycophenolate mofetil (MMF) in inducing remission in treatment-naive patients with autoimmune hepatitis (AIH). The main questions it aims to answer are:

Does MMF combined with prednisolone lead to higher remission rates compared to AZA with prednisolone after 24 weeks? Is MMF associated with fewer adverse events than AZA in these patients? Researchers will compare two treatment arms (MMF vs. AZA) to see if MMF leads to improved remission rates and safety outcomes.

Primary Outcome Measure:

Biochemical remission: The primary outcome is the normalization of liver enzymes (AST, ALT) and IgG levels at 24 weeks.

Secondary Outcome Measures:

Safety and adverse events: Monitoring and comparing the incidence and severity of side effects between the two groups.

Treatment adherence: Evaluating how well patients stick to their assigned treatment regimens.

Improvement in quality of life: Assessing changes in the patient's quality of life using validated questionnaires.

Reversal of fibrosis: Measured by liver stiffness using Fibroscan, aiming for no progression of fibrosis.

Participants will:

Receive either MMF or AZA, alongside a tapering dose of prednisolone. Be monitored regularly through clinic visits, laboratory tests, and safety assessments to track remission and any adverse events.

DETAILED DESCRIPTION:
This clinical trial aims to compare the efficacy and safety of azathioprine (AZA) versus mycophenolate mofetil (MMF) in inducing remission in treatment-naive patients with autoimmune hepatitis (AIH). Autoimmune hepatitis is a chronic liver disease characterized by immune-mediated liver inflammation, leading to liver damage, cirrhosis, or liver failure if untreated.

The study will be conducted at the Institute of Liver and Biliary Sciences (ILBS), where eligible patients with AIH will be randomly assigned to one of two treatment groups:

AZA Group: Patients will receive azathioprine at an initial dose of 50 mg/day, increased to 100 mg/day after two weeks, combined with a tapering dose of prednisolone.

MMF Group: Patients will receive mycophenolate mofetil at an initial dose of 1,000 mg/day, increased to 2,000 mg/day after two weeks, along with a tapering dose of prednisolone.

The trial will enroll 108 patients and follow a double-blind, randomized controlled design. The primary endpoint is achieving biochemical remission within 24 weeks, defined by normalizing liver enzymes (AST, ALT) and IgG levels. Secondary endpoints include safety, tolerability, treatment adherence, quality of life, and the prevention or reversal of liver fibrosis (as measured by Fibroscan).

The trial's expected duration is one year, with follow-up visits every 4 weeks to monitor patient progress and adverse events. All necessary tests and treatments will follow institutional protocols without additional cost to participants.

This study is essential to address the current gaps in AIH treatment, offering critical evidence to guide future clinical decisions on the use of MMF versus AZA for remission induction in AIH.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis: Confirmed diagnosis of autoimmune hepatitis (AIH) based on clinical, biochemical, and histological findings.

Biochemical markers: Elevated liver enzymes, specifically AST and ALT, indicating liver inflammation.

Treatment-naive: Patients must be treatment-naive, meaning they have not received prior immunosuppressive therapy for AIH.

Willingness to participate: Patients must provide informed consent and be willing to comply with all study-related procedures and follow-ups. -

Exclusion Criteria:

* Acute liver failure: Patients presenting with acute liver failure at baseline will be excluded.

Other liver diseases: Co-existing liver conditions such as hepatitis B, hepatitis C, primary biliary cholangitis (PBC), primary sclerosing cholangitis (PSC), or any alcohol-induced liver disease will lead to exclusion.

Low blood counts: Patients with a platelet count less than 50,000/mm³ or total leukocyte count (TLC) less than 3,000/mm³ will not be eligible.

Previous treatment: Patients who have already received immunosuppressive or disease-modifying therapy for AIH or related conditions.

Pregnancy or lactation: Pregnant or lactating women will be excluded to avoid potential risks to the mother or fetus.

Hepatocellular carcinoma (HCC) or malignancy: Any patients with evidence of hepatocellular carcinoma or other active malignancies.

Medication allergies: Patients with known allergies to azathioprine, mycophenolate mofetil (MMF), or prednisolone will be excluded.

Non-consent: Patients who are not willing to participate in the study or unable to provide informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Biochemical Remission at 24 Weeks | 24 weeks
  Definition: Normalization of liver enzymes (ALT, AST) and immunoglobulin G (IgG) levels.
  Time Frame: Measured at 24 weeks of treatment. Purpose: To evaluate the effectiveness of mycophenolate mofetil (MMF) versus azathioprine (AZA) in achieving biochemical remission in treatment-naive autoimmune hepatitis (AIH) patients.

SECONDARY OUTCOMES:
Incidence and Severity of Adverse Events | 24 weeks.
  Definition: Number and severity (mild, moderate, or severe) of adverse events related to the treatment.
  Time Frame: Assessed at each follow-up visit (every 4 weeks) during the 24-week treatment period.
  Purpose: To compare the safety profiles of MMF and AZA.
Treatment Adherence | 24 weeks.
  Definition: Percentage of participants who complete the 24-week treatment without discontinuation due to adverse events or non-compliance.
  Time Frame: Measured throughout the 24-week period. Purpose: To assess patient adherence to treatment protocols in both groups.
Quality of Life Improvement | 24 weeks.
  Definition: Change in the quality of life score based on a validated patient-reported outcome questionnaire, SF-36, and CLDQ.
  Time Frame: Measured at baseline and 24 weeks. Purpose: To determine whether improvements in liver function correlate with better quality of life
Change in Liver Fibrosis | 24 weeks.
  Definition: Change in liver fibrosis stage, measured by Fibroscan. Time Frame: Measured at baseline and 24 weeks. Purpose: To evaluate if either treatment leads to a reduction in liver fibrosis or prevents its progression.

IPD SHARING:
Plan to Share IPD: No
Investigators currently do not plan to share individual participant data (IPD) from this study. The decision is based on considerations of patient privacy, confidentiality concerns, and the lack of a data-sharing infrastructure. While the aggregated study results will be published and made publicly available, sharing individual-level data could pose risks related to identifying participants. Therefore, IPD will not be shared beyond what is required for regulatory purposes.

REFERENCES:
- [Background] Snijders RJALM, Stoelinga AEC, Gevers TJG, Pape S, Biewenga M, Tushuizen ME, Verdonk RC, de Jonge HJM, Vrolijk JM, Bakker SF, Vanwolleghem T, de Boer YS, Baven Pronk MAMC, Beuers U, van der Meer AJ, Gerven NMFV, Sijtsma MGM, van Eijck BC, van IJzendoorn MC, van Herwaarden M, van den Brand FF, Korkmaz KS, van den Berg AP, Guichelaar MMJ, Levens AD, van Hoek B, Drenth JPH; Dutch Autoimmune Hepatitis Working Group. An open-label randomised-controlled trial of azathioprine vs. mycophenolate mofetil for the induction of remission in treatment-naive autoimmune hepatitis. J Hepatol. 2024 Apr;80(4):576-585. doi: 10.1016/j.jhep.2023.11.032. Epub 2023 Dec 14. PMID 38101756
- [Background] Santiago P, Schwartz I, Tamariz L, Levy C. Systematic review with meta-analysis: mycophenolate mofetil as a second-line therapy for autoimmune hepatitis. Aliment Pharmacol Ther. 2019 Apr;49(7):830-839. doi: 10.1111/apt.15157. Epub 2019 Feb 13. PMID 30761563
- [Background] Manns MP, Woynarowski M, Kreisel W, Lurie Y, Rust C, Zuckerman E, Bahr MJ, Gunther R, Hultcrantz RW, Spengler U, Lohse AW, Szalay F, Farkkila M, Prols M, Strassburg CP; European AIH-BUC-Study Group. Budesonide induces remission more effectively than prednisone in a controlled trial of patients with autoimmune hepatitis. Gastroenterology. 2010 Oct;139(4):1198-206. doi: 10.1053/j.gastro.2010.06.046. Epub 2010 Jun 22. PMID 20600032
- [Background] Manns MP, Czaja AJ, Gorham JD, Krawitt EL, Mieli-Vergani G, Vergani D, Vierling JM; American Association for the Study of Liver Diseases. Diagnosis and management of autoimmune hepatitis. Hepatology. 2010 Jun;51(6):2193-213. doi: 10.1002/hep.23584. No abstract available. PMID 20513004
- [Background] Czaja AJ. Current and future treatments of autoimmune hepatitis. Expert Rev Gastroenterol Hepatol. 2009 Jun;3(3):269-91. doi: 10.1586/egh.09.15. PMID 19485809
- [Background] Terziroli Beretta-Piccoli B, Mieli-Vergani G, Vergani D. Autoimmune hepatitis: Standard treatment and systematic review of alternative treatments. World J Gastroenterol. 2017 Sep 7;23(33):6030-6048. doi: 10.3748/wjg.v23.i33.6030. PMID 28970719
- [Background] Sarin SK, Kumar M, Lau GK, Abbas Z, Chan HL, Chen CJ, Chen DS, Chen HL, Chen PJ, Chien RN, Dokmeci AK, Gane E, Hou JL, Jafri W, Jia J, Kim JH, Lai CL, Lee HC, Lim SG, Liu CJ, Locarnini S, Al Mahtab M, Mohamed R, Omata M, Park J, Piratvisuth T, Sharma BC, Sollano J, Wang FS, Wei L, Yuen MF, Zheng SS, Kao JH. Asian-Pacific clinical practice guidelines on the management of hepatitis B: a 2015 update. Hepatol Int. 2016 Jan;10(1):1-98. doi: 10.1007/s12072-015-9675-4. Epub 2015 Nov 13. PMID 26563120
- [Background] Makol A, Watt KD, Chowdhary VR. Autoimmune hepatitis: a review of current diagnosis and treatment. Hepat Res Treat. 2011;2011:390916. doi: 10.1155/2011/390916. Epub 2011 May 15. PMID 21760995
- [Background] Czaja AJ, Freese DK; American Association for the Study of Liver Disease. Diagnosis and treatment of autoimmune hepatitis. Hepatology. 2002 Aug;36(2):479-97. doi: 10.1053/jhep.2002.34944. No abstract available. PMID 12143059